CLINICAL TRIAL: NCT03649282
Title: Comparisons of the Dynamic of the Cardiorespiratory System Behavior of Extreme Preterm Infants Receiving Nasal CPAP or High Flow Nasal Cannula During the Immediate Post-extubation Period
Brief Title: HFNC and NCPAP in Extremely Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guilherme Sant'Anna, MD (Other)
Responsible Party: Sponsor-Investigator, Guilherme Sant'Anna, MD, Associate Professor, Department of Paediatrics, McGill University Health Center, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12-342-PED
Record Dates: First submitted 2018-08-21; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Extreme Prematurity
Keywords: NCPAP; HFNC; Preterm infants; Cardiorespiratory behaviour; Non-invasive respiratory support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC/NCPAP (Experimental): HFNC will be provided for 45 minutes followed by NCPAP for 45 minutes. Cardiorespiratory signals including electrocardiogram (ECG), respiratory inductive plethysmography (RIP), oxygen saturation (SpO2) and Pulse rate will be recorded continuously during the interventions and analyzed offline.
  Interventions: Other: HFNC; Other: NCPAP
- NCPAP/HFNC (Experimental): NCPAP will be provided for 45 minutes followed by HFNC for 45 minutes. Cardiorespiratory signals including electrocardiogram (ECG), respiratory inductive plethysmography (RIP), oxygen saturation (SpO2) and Pulse rate will be recorded continuously during the interventions and analyzed offline.
  Interventions: Other: HFNC; Other: NCPAP

INTERVENTIONS:
Other: HFNC — HFNC therapy will be delivered with a system that provides heated, humidified high flow of gas through a tube that maintains the temperature and humidification. This intervention will involve the delivery of gas (air/oxygen) at a high flow rate, using an adequate nasal cannulae size and a cannula/nostril diameter ratio between 0.5-0.8.
Other: NCPAP — NCPAP will be provided as either bubble CPAP or through a ventilator, and will deliver a regulated pressure of gas (air/oxygen) to the patient through infant binasal prongs as interface. Nasal prong sizes will be chosen according to manufacturer recommendations.

SUMMARY:
To avoid or decrease the rate of complications in preterm infants after disconnection from a mechanical ventilation (extubation), non-invasive respiratory support is routinely used. While infants are most commonly extubated to nasal continuous positive airway pressure (NCPAP), high flow nasal cannula (HFNC) has emerged as an attractive alternative. However, research regarding the safety and efficacy of HFNC in the most extreme preterm infants is limited. Therefore, we hypothesize that immediately after extubation, measures of heart rate and respiratory behavior may be useful to investigate for any differences between HFNC and NCPAP.

DETAILED DESCRIPTION:
Infants will be studied 30 min after extubation on both modes of support, provided in a random order. A transition period of 15 min between modes will be given. For each mode, recordings will be performed for 40 minutes. Analysis of these recordings will be done off line.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weight ≤ 1250 grams
* Infants that have been mechanically ventilated and undergoing their first elective extubation attempt

Exclusion Criteria:

* Major congenital anomalies, neuromuscular disease, hemodynamic instability (use of vasopressors or hypotension).
* Infants reintubated before initiation or during data collection.
* Parental/legal guardian consent not obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Differences on Heart Rate Variability in extremely preterm infants receiving HFNC and NCPAP | Immediate post-extubation period
  Cardiac signals from the electrocardiogram will be continuously measured throughout the recordings. Analysis of these signals will be performed offline to calculate heart rate variability using linear and nonlinear methods.
Differences on Respiratory Variability in extremely preterm infants receiving HFNC and NCPAP | Immediate post-extubation period
  Respiratory variability will be calculated by using analysis of respiratory inductive pletysmography signals from the recordings during HFNC and NCPAP. Desaturation events will also be calculated from these recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Sant'Anna, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided